Quantitative Assessment of Painful Diabetic Peripheral Neuropathy after High Frequency Spinal Cord Stimulation: (QUANT)

HF10 Study

NCT # NCT03769675

27FEB2020



# **General Study Information**

Principal Investigator: Narayan R. Kissoon, MD

Co-Investigators:

Study Title: Quantitative Assessment of Painful Diabetic Peripheral Neuropathy after High Frequency Spinal

Cord Stimulation: (QUANT) HF10 Study

Protocol version number and date: ver. 5 27FEB2020

### **Research Ouestion and Aims**

Hypothesis: Painful lower extremity diabetic peripheral neuropathy (DPN) patients treated with high frequency spinal cord stimulation (HF10 SCS) will have improvements in lower extremity peripheral nerve function.

Aims, purpose, or objectives:

- 1. To determine if patients with DPN have improvements on sensory examination by assessing both small and large fiber modalities after being treated with HF10.
- 2. To determine if patients with DPN have improvements in small fiber nerve function after being treated with HF10 SCS as measured by the quantitative axon reflex sweat test (Q-SWEAT).
- 3. To determine if large fiber nerve function improves after being treated with HF10 SCS as measured by Nerve Conduction Studies of the lower extremities.
- 4. To determine if lower extremity perfusion improves after being treated with HF 10 SCS as measured by Laser Doppler flowmetry.

Background (*Include relevant experience*, gaps in current knowledge, preliminary data, etc.):

Spinal cord stimulation (SCS) has been shown to be effective and is an FDA approved treatment for neuropathic pain of the extremities.<sup>1,2</sup> Randomized trials have demonstrated efficacy in providing pain relief using SCS in patients with neuropathic pain related to diabetic peripheral neuropathy and is an FDA approved treatment for intractable pain related to diabetic peripheral neuropathy.<sup>3-5</sup> Length dependent distal symmetric peripheral polyneuropathy is the most common form of diabetic neuropathy and the pathogenesis is related to vascular (endothelial dysfunction with microvascular ischemia) and metabolic factors (hyperglycemia resulting in oxidative stress).<sup>6-12</sup> These factors lead to progressive neuronal degeneration with the distribution and morphology of fiber loss suggesting ischemia, which is not similar to other diffuse metabolic diseases.<sup>13-19</sup> Vascular physiologic changes such as a reduction of endoneurial oxygen tension has been observed in patients with advanced diabetic polyneuropathy and differences were found between painful and painless diabetic peripheral neuropathy.<sup>20, 21</sup> Animal models of DPN have demonstrated spinally mediated hyperalgesia and allodynia.<sup>22</sup> Pain relief with SCS has been shown to correlate with levels of various neurotrophic factors in the cerebrospinal fluid (CSF).<sup>23, 24</sup>



Growing evidence supports the use of SCS in the treatment of pain-related ischemia with approval in Europe for treatment of refractory angina pectoris and critical limb ischemia.<sup>25</sup> A study by Jivegard et al demonstrated significant pain relief at 18 months for patients with nonsurgical critical limb ischemia when treated with SCS and showed lower amputation rates when excluding patients with arterial hypertension.<sup>26</sup> A study by Broseta et al had shown better outcomes with SCS for critical limb ischemia in patients without hypertension when compared to patients with hypertension.<sup>26, 27</sup> In addition, patients with critical limb ischemia treated with SCS had poorer outcomes with a baseline foot transcutaneous oxygen (TcPO2) < 10 mmHg and clinical improvement coincided with an increase in TcPO2.<sup>28, 29</sup> Other randomized trials not taking into account TcPO2 and history of hypertension did not show any difference between SCS with medical management and medical management alone.<sup>30, 31</sup> A meta-analysis pooled from these prior randomized controlled trials (RCTs) demonstrated significant limb salvage benefit suggesting the individual RCTs were underpowered.<sup>25, 31</sup> Several studies suggest a correlation of pain relief with increased blood perfusion.<sup>32, 33</sup>

In animal models with vasospasm, SCS has been shown to reduce peripheral ischemia. <sup>34,35</sup> The potential improvement in extremity perfusion is believed to result from two mechanisms. <sup>36-39</sup> First, SCS attenuates sympathetic outflow resulting in decreased vascular resistance and increased peripheral blood flow. <sup>36,38,40</sup> Alternatively, SCS can lead to alterations in the ERK and AKT signaling pathways along with GABA release in the grey matter of the spinal cord that results in antidromic activation of primary afferent fibers leading to peripheral vasodilation. <sup>38,41-43</sup> These changes in primary afferent activity are mediated by CGRP release and TRPV1 containing sensory neurons, which can result in nitric oxide-induced endothelium dependent vasodilation. <sup>44-47</sup> In animal models of diabetes, SCS has been shown to increase peripheral blood flow. <sup>48</sup> However, the vasodilatory response was attenuated and thought to be related to the extent of peripheral nerve and autonomic dysfunction. <sup>39,48</sup> The vasodilatory response from SCS appears to be dose dependent with high frequency SCS demonstrating greater increases in cutaneous blood flow when compared to lower frequencies. <sup>36</sup>

In patients with diabetes and critical limb ischemia +/- diabetic neuropathy, improvements in pain relief correlated with increases in peripheral blood flow. <sup>49-51</sup> In patients with diabetes and critical limb ischemia, the severity of autonomic neuropathy was inversely related to the success of SCS therapy (both limb salvage and pain relief), independent of the stage of the peripheral artery disease. <sup>52</sup> In a small case series by de Vos et al 2009, a group of patients with DPN observed significant pain relief, but only a non-significant trend of increased perfusion was seen at 6 months when compared to baseline. <sup>53</sup>

In animal models, SCS has been shown to demonstrate improvements in neurological examination as demonstrated by mechanical withdrawal thresholds (marker of allodynia) and compression withdrawal thresholds (marker of hyperalgesia).<sup>37, 54</sup> These improvements were frequency dependent with changes during treatment using low frequency SCS likely a result of supraspinal mechanisms and changes during higher frequency SCS likely as a result of spinal mechanisms.<sup>54, 55</sup> In a diabetic animal model, high frequency SCS resulted in a delayed effect on pain related behavioral outcome in chronic DPN (mechanical withdrawal thresholds).<sup>37</sup>

HF10 SCS is an FDA approved treatment that has been shown to be superior to traditional lower frequency SCS in the management of chronic back pain and neuropathic lower extremity pain. Freliminary data has C:\Users\mrb4413\Downloads\QUANTHF10 ver5 27FEB2020 clean (2).doc

Page 2 of 14



suggested that treatment of chronic intractable pain related to peripheral polyneuropathy with HF10 SCS also resulted in improvements on neurological examination (predominantly sensory modalities).<sup>57</sup>

Our hypothesis is that patients with painful DPN will have improvements in sensory examination and the improvements will predominantly be in small fiber nerve function. In addition, these improvements may be objectively assessed with small fiber sudomotor testing (Q-SWEAT) as patients with length dependent diabetic peripheral neuropathy have been shown to have sudomotor dysfunction along with progressive sweat gland dennervation. The changes in Q-SWEAT will be an objective marker of small fiber nerve function and the proposed mechanism is through increases in perfusion of the peripheral nerves secondary to vasodilation induced by high frequency spinal cord stimulation. As the HF10 SCS leads are placed at the level of the thoracic segments, it is unlikely to result in any improvements in hand symptoms. Also, SCS would be unlikely to improve upper extremity symptoms in DPN are usually related to superimposed mononeuropathies (median neuropathy at the wrist or ulnar neuropathy at the elbow). 60

Patients with DPN frequently have large nerve fiber involvement as well as the small nerve fiber involvement that will be assessed with Q-SWEAT. Large nerve fiber function can be assessed with nerve conduction studies.

The proposed improvements in peripheral nerve function may occur in both an immediate (days to months) and delayed (months to years) response. Some of the more proximal nerve fibers may be in an area of penumbra where chronic neuropraxia (dysfunctional but still intact) is causing the impairments. With improved perfusion of these fibers, recovery of function may happen more quickly (days to months). In the more distal nerves fibers, the deficits are more likely related to chronic axonotmesis (axonal damage with nerves intact) or neuronotmesis (both axonal and nerve damage), which would likely take more reperfusion time to demonstrate improvements (months to years) with deficits related to axonotmesis. The pain improvement effects of HF10 SCS are sustained with long term data of success with HF10 SCS being demonstrated up to 24 months.<sup>61</sup>

## **Study Design and Methods**

**Methods:** *Describe, in detail, the research activities that will be conducted under this protocol:* 

Patients with intractable neuropathic lower extremity pain related to DPN that fulfill inclusion and exclusion criteria (see below) will be considered for participation in this prospective feasibility study. Baseline testing will be performed to exclude confounding factors that may affect outcomes (figure). All patients that are candidates for SCS undergo a spinal cord stimulation trial as part of standard clinical care with all of the FDA approved indications. If the patient is deemed a candidate and complying with this standard clinical practice, the patient will undergo a HF10 SCS (Nevro Senza®) trial lasting up to 14 days with an external stimulator to determine short term response. For Patients with 40% or greater pain reduction from baseline will be eligible to proceed to permanent implantation. Fatients with HF10 SCS will receive 30 µs pulses delivered at 10,000 Hz with amplitude adjusted to optimal analgesic response. Programming will occur postoperatively and as needed based on patient feedback in standard clinic visits. At 6 month follow-up, paresthesia mapping will be performed during the programming visit in which the subthreshold SCS will be temporary increased during a 10 minute protocol to a perceived level to determine the dermatomal stimulation pattern with the SCS lead placement.



# Implant Procedures

The SCS implant will follow standard clinical practice for these FDA approved indications. Two percutaneous leads will be placed in the posterior spinal epidural space under radiographic guidance and attached to either an external stimulator (trial phase) or a subcutaneously implanted impulse generator (IPG). The distal tip of one lead will be placed at the top of the T8 vertebral body and the second lead tip will be placed at the mid T9 vertebral level for maximal electrode coverage at the T9/T10 junction. A subcutaneous pocket will be created using standard surgical techniques for placement of an IPG. The leads, anchored to the supraspinous fascia, will be tunneled to the pocket site and connected to the IPG. Intraoperative impedance testing will be performed to ensure electrical integrity.

#### Outcome Assessments

Adverse events will be monitored throughout the study (e.g. infection, lead migration). Lead migration will be defined as loss of efficacy that could not be remedied by reprogramming and confirmed radiologically.<sup>56</sup> Baseline testing will be performed either prior to SCS trial or a minimum of two weeks following removal of SCS trial leads and prior to SCS implant. During outcome assessments, the spinal cord stimulator will remain active and any medications that can impact autonomic testing will be discontinued prior to each test. Assessments of pain will be made with the numeric rating scale (NRS) for each of the time points. The patient will be contacted at 5 and 11 months to set up in-person assessment appointments. At this time, the NRS will be used. If the NRS is >3 the principal investigator will be notified and the patient will have an appointment for a SCS assessment prior to the 6 and 12 month assessment. Neuropathic symptoms will be monitored with the Neuropathy Symptoms and Change (NSC) scale at 6 months and 12 months to assess impact on neuropathic pain (figure). <sup>62</sup> Patient Health Questionnaire (PHQ9) will be assessed at baseline, 6 months and 12 months to monitor for the presence and severity of depression. A body mass index (BMI) and Hemoglobin A1C (HgA1C) will be done at baseline and at 12 months. The presence of allodynia and/or hyperalgesia will be monitored throughout the course of the study with the modified Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS).<sup>63</sup> Small fiber sudomotor function with Q-SWEAT will be assessed periodically during the study (baseline, 6 months, and 12 months) (figure). 28, 53, 58, 59, 64, 65

Gross neurologic function will be assessed by a board certified neurologist at baseline, 6 months, and 12 months, and the neuropathy impairment score (NIS) of the lower limbs with lower limb function test (LLF) will be calculated for an objective comparative assessment. EMG will be performed at baseline (partly to exclude mimickers of DPN) and at 12 months to compare nerve conduction studies (NCS) for an objective assessment of large fiber nerve function(figure). Only the NCS of the lower limb will be performed with the EMG at 12 months (no needle EMG will be performed at 12 months). The Oswestry Disability Index (ODI) will be used as a gross functional assessment at each of the time points.

**Resources:** Describe the available resources to conduct the research (personnel, time, facilities, mentor commitment, etc.):

- 1. Clinical research coordinator to aid in implementation of the study
- 2. Periodic testing (Q-SWEAT and Laser Doppler flowmetry) will be performed in the Clinical Research Unit (CRU)



| (1a) This is a multisite study involving Mayo Clinic and non Mayo Clinic sites. When check | ked, describe in |
|---|---|
| detail the research procedures or activities that will be conducted by Mayo Clinic study staff. | |
| [16] Mayo Clinic study staff will be engaged in research activity at a non Mayo Clinic site. | When checked, |
| provide a detailed description of the activity that will be conducted by Mayo Clinic study staff. | |

# **Subject Information**

Target accrual is the proposed total number of subjects to be included in this study at Mayo Clinic. A "Subject" may include medical records, images, or specimens generated at Mayo Clinic and/or received from external sources.

Target accrual: 20 patients over the course of a 2 year enrollment period (3 years in total for completion of study).

Subject population (children, adults, groups): Patients with the FDA approved indication of medically intractable painful DPN age 18 and over that are appropriate surgical candidates and without severe autonomic neuropathy or psychiatric comorbidity that would preclude SCS implant.

### Inclusion Criteria:

- $\geq$  18 years of age
- Type 2 diabetes mellitus
- Refractory predominantly lower extremity neuropathic pain for > 1 year
- Presence of length dependent peripheral neuropathy on sudomotor testing (Q-SWEAT)
- Completed spinal cord stimulation trial with 40% or greater pain reduction from baseline
- Failed medication trials or contraindication to gabapentinoid medications (gabapentin, pregabalin) and/or serotonin/norepinephrine reuptake inhibitors (tricyclic antidepressant (TCA) or duloxetine or venlafaxine)
- Average pain score on a numeric rating scale of  $\geq 5$  (with 0 representing no pain and 10 the worst pain imaginable)
- Appropriate surgical candidate for SCS<sup>56</sup>

## **Exclusion Criteria:**

- Severe Autonomic Neuropathy as measured by the composite autonomic scoring scale (10 point scale) with a score  $\geq 7^{52, 64}$
- History of sympathectomy<sup>52</sup>
- Uncontrolled arterial hypertension (Systolic Blood Pressure >160)<sup>26, 27</sup>
- Baseline Foot TcPO2 < 10 mmHg to exclude patients with severe peripheral arterial disease<sup>28, 29</sup>
- Hemoglobin A1c >  $8\%^{68, 69}$
- Stable opioid regimen with oral morphine equivalent  $\geq 100 \text{ mg/day}^{70}$
- Alternative principle cause for peripheral neuropathy or lower extremity neuropathic pain
- Disruptive psychiatric disorder (screened for during preoperative psychiatric evaluation)<sup>56</sup>
- Pending litigations<sup>56</sup>



- Women of child bearing potential unwilling to use contraception or found to be pregnant as part of perioperative screening
- Patients unable to hold medications that would impact autonomic testing

## **Research Activity**

Check all that apply and complete the appropriate sections as instructed.

| CII | check all that apply and complete the appropriate sections as instructed. |
|---|---|
| 1. | Drug & Device: Drugs for which an investigational new drug application is not required. Device for which (i) an investigational device exemption application is not required; or the medical device is cleared/approved for marketing and being used in accordance with its cleared/approved labeling. (Specify in the Methods section) |
| 2. | ☐ <b>Blood</b> : Collection of blood samples by finger stick, heel stick, ear stick, or venipuncture. |
| 3. | Biological specimens other than blood: Prospective collection of human biological specimens by noninvasive means that may include: urine, sweat, saliva, buccal scraping, oral/anal/vaginal swab, sputum, hair and nail clippings, etc. |
| 4. | Tests & Procedures: Collection of data through noninvasive tests and procedures routinely employed in clinical practice that may include: MRI, surface EEG, echo, ultrasound, moderate exercise, muscular strength & flexibility testing, biometrics, cognition testing, eye exam, etc. (Specify in the Methods section) |
| 5. | <b>Data</b> (medical record, images, or specimens): Research involving use of existing and/or prospectively collected data. |
| 6. | ☐ <b>Digital Record</b> : Collection of electronic data from voice, video, digital, or image recording. (Specify in the Methods section) |
| 7. | ☐ Survey, Interview, Focus Group: Research on individual or group characteristics or behavior, survey, interview, oral history, focus group, program evaluation, etc. (Specify in the Methods section) |
| <br>inv | NIH has issued a Certificate of Confidentiality (COC). When checked, provide the institution and restigator named on the COC and explain why one was requested. |
| | Biospecimens – Categories 2 and 3 |

- (2) Collection of blood samples. When multiple groups are involved copy and paste the appropriate section below for example repeat section b when drawing blood from children and adults with cancer.
  - a. **From healthy, non-pregnant, adult subjects who weigh at least 110 pounds**. For a minimal risk application, the amount of blood drawn from these subjects may not exceed 550ml in an 8 week period and collection may not occur more frequently than 2 times per week.



| Volume per blood draw:ml Frequency of blood draw (e.g. single draw, time(s) per week, per year, etc.) |
|---|
| b. From other adults and children considering age, weight, and health of subject. For a minimal risk application, the amount of blood drawn from these subjects may not exceed the lesser of 50 ml or 3 ml per kg in an 8 week period, and collection may not occur more frequently than 2 times per week. Volume per blood draw:ml Frequency of blood draw (e.g. single draw, time(s) per week, per year, etc.) |
| (3) Prospective collection of biological specimens other than blood: |
| Review of medical records, images, specimens – Category 5 |
| For review of existing data: provide a date range or an end date for when the data was generated. The end date can be the date this application was submitted to the IRB. Example: 01/01/1999 to 12/31/2015 or all records through mm/dd/yyyy. |
| Date Range: 01/01/2015 to 6/30/2022 |
| Check all that apply (data includes medical records, images, specimens). |
| (5a) Only data that exists before the IRB submission date will be collected. |
| (5b) The study involves data that exist at the time of IRB submission <b>and</b> data that will be generated after IRB submission. Include this activity in the <u>Methods</u> section. |
| <ul> <li>The study plans to conduct a retrospective chart review and ask subjects to complete a questionnaire.</li> <li>The study plans to include subjects previously diagnosed with a specific disease and add newly diagnosed subjects in the future.</li> <li>(5c) The study will use data that have been collected under another IRB protocol. Include in the Methods section and enter the IRB number from which the research material will be obtained. When appropriate, note when subjects have provided consent for future use of their data and/or specimens as described in this protocol.</li> </ul> |
| Enter one IRB number per line, add more lines as needed |
| ☐ Data ☐ Specimens ☐ Data & Specimens |
| ☐ Data ☐ Specimens ☐ Data & Specimens |
| ☐ Data ☐ Specimens ☐ Data & Specimens |



| (5d) This study will obtain data generated from other sources. Examples may include receiving data from participating sites or an external collaborator, accessing an external database or registry, etc. Explain the source and how the data will be used in the Methods section. |
|---|
| (6) Video audio recording: Describe the plan to maintain subject privacy and data confidentiality, transcription, store or destroy, etc. |

## HIPAA Identifiers and Protected Health Information (PHI)

Protected health information is medical data that can be linked to the subject directly or through a combination of indirect identifiers.

Recording identifiers (including a code) during the conduct of the study allows you to return to the medical record or data source to delete duplicate subjects, check a missing or questionable entry, add new data points, etc. De-identified data is medical information that has been stripped of <u>all</u> HIPAA identifiers so that it cannot be linked back to the subject. De-identified data is **rarely** used in the conduct of a research study involving a chart review.

Review the list of subject identifiers below and, if applicable, check the box next to each HIPAA identifier being recorded at the time of data collection or abstraction. Identifiers apply to any subject enrolled in the study including Mayo Clinic staff, patients and their relatives and household members.

**Internal** refers to the subject's identifier that will be recorded at Mayo Clinic by the study staff. **External** refers to the subject's identifier that will be shared outside of Mayo Clinic.

| Check all that apply: | INTERNAL | EXTERNAL |
|---|---|---|
| Name | X | |
| Mayo Clinic medical record or patient registration number, lab accession, specimen or radiologic image number | X | |
| Subject ID, subject code or any other person-specific unique identifying number, characteristic or code that can link the subject to their medical data | X | |
| Dates: All elements of dates [month, day, and year] directly related to an individual, their birth date, date of death, date of diagnosis, etc. | X | |
| <b>Note:</b> Recording a year only is not a unique identifier. | | |
| Social Security number | X | |
| Medical device identifiers and serial numbers | X | |
| Biometric identifiers, including finger and voice prints, full face photographic images and any comparable images | | |
| Web Universal Resource Locators (URLs), Internet Protocol (IP) address numbers, email address | | |
| Street address, city, county, precinct, zip code, and their equivalent geocodes | | |



| Phone or fax numbers | | |
|---|---|---|
| Account, member, certificate or professional license numbers, health | | |
| beneficiary numbers | | |
| Vehicle identifiers and serial numbers, including license plate numbers | | |
| Check 'None' when none of the identifiers listed above will be recorded, | None | None |
| maintained, or shared during the conduct of this study. (exempt category 4) | None | None |

## Data Analysis

Power analyses and study endpoints are not required for minimal risk research, pilot or feasibility studies.

No statistical information. *If checked, please explain*: feasibility study.

#### Power Statement:

This is a feasibility study and so a power analysis was not performed.

Data Analysis Plan: Demographic data will be reported with descriptive statistics, including means with SD's for continuous data and percentages and counts for categorical data. Assuming a normal distribution, two-sided paired t tests and analysis of covariance (ANCOVA) will be used to compare means in VAS/NRS pain scores, NSC, ODI, NIS, LLF, and S-LANSS scores at the corresponding time points as the primary endpoints(figure). In addition, two-sided paired t tests and analysis of covariance (ANCOVA) will be used to compare means for amplitudes (mA) and conduction velocity (m/s) on NCS with EMG at baseline and 12 months post-implant. The secondary endpoints will be assessed with two-sided paired t tests and analysis of covariance (ANCOVA) for latency (min) and sweat output ( $\mu$ L/cm²) on Q-SWEAT and arbitrary perfusion units on Laser Doppler flowmetry (p.u.) at baseline, 6 months, and 12 months post-implant.

#### Endpoints:

Primary: Changes in VAS/NRS, NSC, ODI, NIS, LLF, and S-LANSS.

Secondary: Changes in latency (min) and sweat output (µL/cm²) on Q-SWEAT, arbitrary perfusion units (p.u.) on Laser Doppler flowmetry, and amplitudes (mA) and conduction velocity (m/s) on NCS when compared to baseline. Changes in BMI, HgA1C and PHQ9 scores when compared to baseline.

**FIGURE** 



# Quantitative Assessment of Painful Diabetic Peripheral Neuropathy after High Frequency Spinal Cord Stimulation: (QUANT) HF10 Study



## **REFERENCES:**

- 1. Kumar K, Taylor RS, Jacques L, et al. Spinal cord stimulation versus conventional medical management for neuropathic pain: a multicentre randomised controlled trial in patients with failed back surgery syndrome. Pain 2007;132:179-188.
- 2. Kemler MA, Barendse GA, van Kleef M, et al. Spinal cord stimulation in patients with chronic reflex sympathetic dystrophy. N Engl J Med 2000;343:618-624.
- 3. Slangen R, Schaper NC, Faber CG, et al. Spinal cord stimulation and pain relief in painful diabetic peripheral neuropathy: a prospective two-center randomized controlled trial. Diabetes Care 2014;37:3016-3024.
- 4. de Vos CC, Meier K, Zaalberg PB, et al. Spinal cord stimulation in patients with painful diabetic neuropathy: a multicentre randomized clinical trial. Pain 2014;155:2426-2431.
- 5. van Beek M, Slangen R, Schaper NC, et al. Sustained Treatment Effect of Spinal Cord Stimulation in Painful Diabetic Peripheral Neuropathy: 24-Month Follow-up of a Prospective Two-Center Randomized Controlled Trial. Diabetes Care 2015;38:e132-134.
- 6. Dyck PJ, Kratz KM, Karnes JL, et al. The prevalence by staged severity of various types of diabetic neuropathy, retinopathy, and nephropathy in a population-based cohort: the Rochester Diabetic Neuropathy Study. Neurology 1993;43:817-824.
- 7. Edwards JL, Vincent AM, Cheng HT, Feldman EL. Diabetic neuropathy: mechanisms to management. Pharmacol Ther 2008;120:1-34.
- 8. Kilo S, Berghoff M, Hilz M, Freeman R. Neural and endothelial control of the microcirculation in diabetic peripheral neuropathy. Neurology 2000;54:1246-1252.



- 9. Tesfamariam B, Brown ML, Cohen RA. Elevated glucose impairs endothelium-dependent relaxation by activating protein kinase C. J Clin Invest 1991;87:1643-1648.
- 10. Roustit M, Loader J, Deusenbery C, Baltzis D, Veves A. Endothelial Dysfunction as a Link Between Cardiovascular Risk Factors and Peripheral Neuropathy in Diabetes. J Clin Endocrinol Metab 2016;101:3401-3408.
- 11. Karasu C, Dewhurst M, Stevens EJ, Tomlinson DR. Effects of anti-oxidant treatment on sciatic nerve dysfunction in streptozotocin-diabetic rats; comparison with essential fatty acids. Diabetologia 1995;38:129-134.
- 12. Pieper GM, Gross GJ. Oxygen free radicals abolish endothelium-dependent relaxation in diabetic rat aorta. Am J Physiol 1988;255:H825-833.
- 13. Partanen J, Niskanen L, Lehtinen J, Mervaala E, Siitonen O, Uusitupa M. Natural history of peripheral neuropathy in patients with non-insulin-dependent diabetes mellitus. N Engl J Med 1995;333:89-94.
- 14. Dyck PJ, Karnes JL, O'Brien P, Okazaki H, Lais A, Engelstad J. The spatial distribution of fiber loss in diabetic polyneuropathy suggests ischemia. Ann Neurol 1986;19:440-449.
- 15. Dyck PJ, Hansen S, Karnes J, et al. Capillary number and percentage closed in human diabetic sural nerve. Proc Natl Acad Sci U S A 1985;82:2513-2517.
- 16. Malik RA, Tesfaye S, Newrick PG, et al. Sural nerve pathology in diabetic patients with minimal but progressive neuropathy. Diabetologia 2005;48:578-585.
- 17. Dyck PJ, Lais A, Karnes JL, O'Brien P, Rizza R. Fiber loss is primary and multifocal in sural nerves in diabetic polyneuropathy. Ann Neurol 1986;19:425-439.
- 18. Vracko R. A comparison of the microvascular lesions in diabetes mellitus with those in normal aging. J Am Geriatr Soc 1982;30:201-205.
- 19. Williams E, Timperley WR, Ward JD, Duckworth T. Electron microscopical studies of vessels in diabetic peripheral neuropathy. J Clin Pathol 1980;33:462-470.
- 20. Newrick PG, Wilson AJ, Jakubowski J, Boulton AJ, Ward JD. Sural nerve oxygen tension in diabetes. Br Med J (Clin Res Ed) 1986;293:1053-1054.
- 21. Eaton SE, Harris ND, Ibrahim S, et al. Increased sural nerve epineurial blood flow in human subjects with painful diabetic neuropathy. Diabetologia 2003;46:934-939.
- 22. Jolivalt CG, Lee CA, Ramos KM, Calcutt NA. Allodynia and hyperalgesia in diabetic rats are mediated by GABA and depletion of spinal potassium-chloride co-transporters. Pain 2008;140:48-57.
- 23. McCarthy KF, Connor TJ, McCrory C. Cerebrospinal fluid levels of vascular endothelial growth factor correlate with reported pain and are reduced by spinal cord stimulation in patients with failed back surgery syndrome. Neuromodulation 2013;16:519-522; discussion 522.
- 24. McCarthy KF, McCrory C. Cerebrospinal fluid levels of glial cell-derived neurotrophic factor correlate with spinal cord stimulation frequency in patients with neuropathic pain: a preliminary report. Spinal Cord 2014;52 Suppl 2:S8-10.
- 25. Song JJ, Popescu A, Bell RL. Present and potential use of spinal cord stimulation to control chronic pain. Pain Physician 2014;17:235-246.
- 26. Jivegard LE, Augustinsson LE, Holm J, Risberg B, Ortenwall P. Effects of spinal cord stimulation (SCS) in patients with inoperable severe lower limb ischaemia: a prospective randomised controlled study. Eur J Vasc Endovasc Surg 1995;9:421-425.
- 27. Broseta J, Barbera J, de Vera JA, et al. Spinal cord stimulation in peripheral arterial disease. A cooperative study. J Neurosurg 1986;64:71-80.
- 28. Claeys LG, Horsch S. Transcutaneous oxygen pressure as predictive parameter for ulcer healing in endstage vascular patients treated with spinal cord stimulation. Int Angiol 1996;15:344-349.



- 29. Claeys LG. Improvement of microcirculatory blood flow under epidural spinal cord stimulation in patients with nonreconstructible peripheral arterial occlusive disease. Artif Organs 1997;21:201-206.
- 30. Klomp HM, Spincemaille GH, Steyerberg EW, Habbema JD, van Urk H. Spinal-cord stimulation in critical limb ischaemia: a randomised trial. ESES Study Group. Lancet 1999;353:1040-1044.
- 31. Ubbink DT, Vermeulen H. Spinal cord stimulation for non-reconstructable chronic critical leg ischaemia. Cochrane Database Syst Rev 2003:CD004001.
- 32. Ubbink DT, Spincemaille GH, Prins MH, Reneman RS, Jacobs MJ. Microcirculatory investigations to determine the effect of spinal cord stimulation for critical leg ischemia: the Dutch multicenter randomized controlled trial. J Vasc Surg 1999;30:236-244.
- 33. Naoum JJ, Arbid EJ. Spinal cord stimulation for chronic limb ischemia. Methodist Debakey Cardiovasc J 2013;9:99-102.
- 34. Linderoth B, Gherardini G, Ren B, Lundeberg T. Severe peripheral ischemia after vasospasm may be prevented by spinal cord stimulation. A preliminary report of a study in a free-flap animal model. Acta Neurochir Suppl 1995;64:101-105.
- 35. Linderoth B, Gherardini G, Ren B, Lundeberg T. Preemptive spinal cord stimulation reduces ischemia in an animal model of vasospasm. Neurosurgery 1995;37:266-271; discussion 271-262.
- 36. Gao J, Wu M, Li L, et al. Effects of spinal cord stimulation with "standard clinical" and higher frequencies on peripheral blood flow in rats. Brain Res 2010;1313:53-61.
- 37. van Beek M, van Kleef M, Linderoth B, van Kuijk SM, Honig WM, Joosten EA. Spinal cord stimulation in experimental chronic painful diabetic polyneuropathy: Delayed effect of High-frequency stimulation. Eur J Pain 2016.
- 38. Linderoth B, Fedorcsak I, Meyerson BA. Peripheral vasodilatation after spinal cord stimulation: animal studies of putative effector mechanisms. Neurosurgery 1991;28:187-195.
- 39. Tanaka S, Barron KW, Chandler MJ, Linderoth B, Foreman RD. Local cooling alters neural mechanisms producing changes in peripheral blood flow by spinal cord stimulation. Auton Neurosci 2003;104:117-127.
- 40. Linderoth B, Herregodts P, Meyerson BA. Sympathetic mediation of peripheral vasodilation induced by spinal cord stimulation: animal studies of the role of cholinergic and adrenergic receptor subtypes. Neurosurgery 1994;35:711-719.
- 41. Wu M, Komori N, Qin C, Farber JP, Linderoth B, Foreman RD. Extracellular signal-regulated kinase (ERK) and protein kinase B (AKT) pathways involved in spinal cord stimulation (SCS)-induced vasodilation. Brain Res 2008;1207:73-83.
- 42. Tanaka S, Komori N, Barron KW, Chandler MJ, Linderoth B, Foreman RD. Mechanisms of sustained cutaneous vasodilation induced by spinal cord stimulation. Auton Neurosci 2004;114:55-60.
- 43. Tanaka S, Barron KW, Chandler MJ, Linderoth B, Foreman RD. Role of primary afferents in spinal cord stimulation-induced vasodilation: characterization of fiber types. Brain Res 2003;959:191-198.
- 44. Wu M, Komori N, Qin C, Farber JP, Linderoth B, Foreman RD. Roles of peripheral terminals of transient receptor potential vanilloid-1 containing sensory fibers in spinal cord stimulation-induced peripheral vasodilation. Brain Res 2007;1156:80-92.
- 45. Wu M, Komori N, Qin C, Farber JP, Linderoth B, Foreman RD. Sensory fibers containing vanilloid receptor-1 (VR-1) mediate spinal cord stimulation-induced vasodilation. Brain Res 2006;1107:177-184.
- 46. Yang X, Farber JP, Wu M, Foreman RD, Qin C. Roles of dorsal column pathway and transient receptor potential vanilloid type 1 in augmentation of cerebral blood flow by upper cervical spinal cord stimulation in rats. Neuroscience 2008;152:950-958.



- 47. Tanaka S, Barron KW, Chandler MJ, Linderoth B, Foreman RD. Low intensity spinal cord stimulation may induce cutaneous vasodilation via CGRP release. Brain Res 2001;896:183-187.
- 48. Wu M, Thorkilsen MM, Qin C, Farber JP, Linderoth B, Foreman RD. Effects of spinal cord stimulation on peripheral blood circulation in rats with streptozotocin-induced diabetes. Neuromodulation 2007;10:216-223.
- 49. Petrakis E, Sciacca V. Prospective study of transcutaneous oxygen tension (TcPO2) measurement in the testing period of spinal cord stimulation in diabetic patients with critical lower limb ischaemia. Int Angiol 2000;19:18-25.
- 50. Petrakis IE, Sciacca V. Epidural spinal cord electrical stimulation in diabetic critical lower limb ischemia. J Diabetes Complications 1999;13:293-299.
- 51. Petrakis IE, Sciacca V. Spinal cord stimulation in diabetic lower limb critical ischaemia: transcutaneous oxygen measurement as predictor for treatment success. Eur J Vasc Endovasc Surg 2000;19:587-592.
- 52. Petrakis IE, Sciacca V. Does autonomic neuropathy influence spinal cord stimulation therapy success in diabetic patients with critical lower limb ischemia? Surg Neurol 2000;53:182-188; discussion 188-189.
- 53. de Vos CC, Rajan V, Steenbergen W, van der Aa HE, Buschman HP. Effect and safety of spinal cord stimulation for treatment of chronic pain caused by diabetic neuropathy. J Diabetes Complications 2009;23:40-45.
- 54. Maeda Y, Wacnik PW, Sluka KA. Low frequencies, but not high frequencies of bi-polar spinal cord stimulation reduce cutaneous and muscle hyperalgesia induced by nerve injury. Pain 2008;138:143-152.
- 55. Maeda Y, Ikeuchi M, Wacnik P, Sluka KA. Increased c-fos immunoreactivity in the spinal cord and brain following spinal cord stimulation is frequency-dependent. Brain Res 2009;1259:40-50.
- 56. Kapural L, Yu C, Doust MW, et al. Novel 10-kHz High-frequency Therapy (HF10 Therapy) Is Superior to Traditional Low-frequency Spinal Cord Stimulation for the Treatment of Chronic Back and Leg Pain: The SENZA-RCT Randomized Controlled Trial. Anesthesiology 2015;123:851-860.
- 57. Galan V CP, Scowcroft J, Li S, Staats P. A prospective clinical trial to assess the feasibility of high frequency spinal cord stimulation (HF-SCS) at 10 kHz in the treatment of chronic intractable pain from peripheral polyneuropathy. 2017.
- 58. Fealey RD, Low PA, Thomas JE. Thermoregulatory sweating abnormalities in diabetes mellitus. Mayo Clin Proc 1989;64:617-628.
- 59. Liu Y, Billiet J, Ebenezer GJ, et al. Factors influencing sweat gland innervation in diabetes. Neurology 2015;84:1652-1659.
- 60. Tracy JA, Dyck PJ. The spectrum of diabetic neuropathies. Phys Med Rehabil Clin N Am 2008;19:1-26, v.
- 61. Kapural L, Yu C, Doust MW, et al. Comparison of 10-kHz High-Frequency and Traditional Low-Frequency Spinal Cord Stimulation for the Treatment of Chronic Back and Leg Pain: 24-Month Results From a Multicenter, Randomized, Controlled Pivotal Trial. Neurosurgery 2016;79:667-677.
- 62. Dyck PJ, Turner DW, Davies JL, et al. Electronic case-report forms of symptoms and impairments of peripheral neuropathy. Can J Neurol Sci 2002;29:258-266.
- 63. Bennett MI, Smith BH, Torrance N, Potter J. The S-LANSS score for identifying pain of predominantly neuropathic origin: validation for use in clinical and postal research. J Pain 2005;6:149-158.
- 64. Low PA. Composite autonomic scoring scale for laboratory quantification of generalized autonomic failure. Mayo Clin Proc 1993;68:748-752.
- 65. Divisova S, Vlckova E, Srotova I, et al. Intraepidermal nerve-fibre density as a biomarker of the course of neuropathy in patients with Type 2 diabetes mellitus. Diabet Med 2016;33:650-654.
- 66. Dyck PJ, Herrmann DN, Staff NP, Dyck PJ. Assessing decreased sensation and increased sensory phenomena in diabetic polyneuropathies. Diabetes 2013;62:3677-3686.



- 67. Dyck PJ, Davies JL, Litchy WJ, O'Brien PC. Longitudinal assessment of diabetic polyneuropathy using a composite score in the Rochester Diabetic Neuropathy Study cohort. Neurology 1997;49:229-239.
- 68. Themistocleous AC, Ramirez JD, Shillo PR, et al. The Pain in Neuropathy Study (PiNS): a cross-sectional observational study determining the somatosensory phenotype of painful and painless diabetic neuropathy. Pain 2016;157:1132-1145.
- 69. van de Poll-Franse LV, Valk GD, Renders CM, Heine RJ, van Eijk JT. Longitudinal assessment of the development of diabetic polyneuropathy and associated risk factors. Diabet Med 2002;19:771-776.
- 70. Low PA. Testing the autonomic nervous system. Semin Neurol 2003;23:407-421.